CLINICAL TRIAL: NCT01008995
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Study Evaluating the Efficacy and Safety of Ustekinumab in the Treatment of Chinese Subjects With Moderate to Severe Plaque-type Psoriasis
Brief Title: A Study of the Safety and Effectiveness of Ustekinumab (Stelara) in Chinese Patients With Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR016318; C0743T23 (Other: Centocor); CR016318 (Other: Centocor)
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Results first posted 2012-09-14 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-10

CONDITIONS: Psoriasis
Keywords: psoriasis; asian patients; Chinese; ustekinumab; CNTO 1275; Stelara
MeSH Terms: conditions — Psoriasis | interventions — Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 001 (Experimental): placebo Subcutaneous injection at Week 0 and 4,ustekinumab 45 mg subcutaneous injection at Week 12 and 16
  Interventions: Drug: placebo; Drug: ustekinumab
- 002 (Experimental): placebo Subcutaneous injection at Week 12,ustekinumab 45 mg subcutaneous injection at Week 0 4 and 16
  Interventions: Drug: placebo; Drug: ustekinumab

INTERVENTIONS:
Drug: placebo — Subcutaneous injection at Week 0 and 4
  Arms: 001
Drug: ustekinumab — 45 mg subcutaneous injection at Week 12 and 16
  Arms: 001
Drug: placebo — Subcutaneous injection at Week 12
  Arms: 002
Drug: ustekinumab — 45 mg subcutaneous injection at Week 0, 4 and 16
  Arms: 002

SUMMARY:
The purpose of this study is to evaluate the efficacy (good or bad effects) and safety of ustekinumab in the treatment of patients with moderate to severe psoriasis in China.

DETAILED DESCRIPTION:
In this study, 220 patients will be divided into two groups randomly (by chance), like flipping a coin. Each group will receive a different treatment. The results for each group are compared to each other. There are 2 treatment groups in this study, Group 1 and Group 2. Group 1 will receive placebo at Weeks 0 and 4, ustekinumab 45 mg at Weeks 12 and 16. Group 2 will receive ustekinumab 45 mg at Weeks 0, 4, and 16 and placebo at Week 12. All patients in the study will eventually receive ustekinumab after Week 12. The patients will be in the study for about 36 weeks, with study visit approximately 10 times. Effectiveness evaluations will be conducted throughout the study and include the Psoriasis Area and Severity Index (PASI), Physician's Global Assessment (PGA) and Dermatology Life Quality Index (DLQI). Safety assessments will also be performed throughout the study and include obtaining and evaluating laboratory tests, vital signs (e.g., blood pressure) and the occurrence and severity of adverse events. GROUP 1: Placebo at Weeks 0 and 4, ustekinumab 45 mg at Weeks 12 and 16. GROUP 2: Ustekinumab 45 mg at Weeks 0, 4, and 16. Placebo at Week 12

ELIGIBILITY:
Inclusion Criteria:

* Must be of Chinese ancestry
* Have had a diagnosis of plaque-type psoriasis at least 6 months prior to study start
* Have plaque-type psoriasis covering at least 10% of total BSA at screening and at the time of study start
* Have a Psoriasis Area and Severity Index (PASI) score of 12 or greater at study start
* Must be candidates for phototherapy or systemic treatment of psoriasis (either naive or history of previous treatment)

Exclusion Criteria:

* Currently have nonplaque forms of psoriasis
* Have current drug-induced psoriasis
* Have used any investigational drug within the previous 4 weeks
* Have used any biologic within the previous 3 months
* Be known to be infected with human immunodeficiency virus (HIV), hepatitis B virus (HBV), hepatitis C virus (HCV), or syphilis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2009-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.
Locations (9):
- China (9):
  - Beijing
  - Chongqing
  - Dalian
  - Guangzhou
  - Hangzhou
  - Nanjing
  - Shanghai
  - Shenyang
  - Xi'an

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo (CP): Controlled period (Week 0-12) - Placebo Group
- Ustekinumab 45 mg (CP): Controlled period (Week 0-12) - Ustekinumab 45 mg Group
- Placebo -> Ustekinumab 45 mg (After CP): After controlled period (Week 12-36) - receiving Placebo at Weeks 0 and 4 -> receiving ustekinumab 45 mg at Week 12 and Week 16
- Ustekinumab 45 mg (After CP): After controlled period (Week 12-36) - receiving ustekinumab 45 mg at Weeks 0 and 4 -> receiving placebo at Week 12 and ustekinumab 45 mg at Week 16
Period: Controlled Period
Arm/Group | Placebo (CP) | Ustekinumab 45 mg (CP) | Placebo -> Ustekinumab 45 mg (After CP) | Ustekinumab 45 mg (After CP)
Started | 162 | 160 | 0 ("0" in column indicates this reporting group is not relevant to Control Period.) | 0 ("0" in column indicates this reporting group is not relevant to Control Period.)
Completed | 159 | 157 | 0 | 0
Not Completed | 3 | 3 | 0 | 0
Not completed — Adverse Event | 1 | 2 | 0 | 0
Not completed — Other | 2 | 1 | 0 | 0
Period: After Controlled Period
Arm/Group | Placebo (CP) | Ustekinumab 45 mg (CP) | Placebo -> Ustekinumab 45 mg (After CP) | Ustekinumab 45 mg (After CP)
Started | 0 ("0" in column indicates this reporting group is not relevant to after Control Period.) | 0 ("0" in column indicates this reporting group is not relevant to after Control Period.) | 158 (1 placebo participant discontinued after completing the CP and did not receive ustekinumab 45 mg.) | 157 (2 participants discontinued in CP, had follow-up, and are among frequent and serious adverse events.)
Completed | 0 | 0 | 156 | 156
Not Completed | 0 | 0 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 1
Not completed — Other | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (CP) | Ustekinumab 45 mg (CP) | Total
Number analyzed (Participants) | 162 | 160 | 322
Age Continuous [Mean (Standard Deviation); unit: years] | 39.2 (12.21) | 40.1 (12.36) | 39.7 (12.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 35 | 74
  Male | 123 | 125 | 248
Region of Enrollment [Number; unit: participants]
  China | 162 | 160 | 322

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients Who Achieved at Least a 75% Improvement in PASI (Psoriasis Area and Severity Index) From Baseline at Week 12.
Description: Scores could range from 0 (mild) to 72 (severe).
Time Frame: Baseline (Week 0) to Week 12
Population: All participants were analyzed according to the treatment group to which they were randomized, regardless of the treatment they actually received.
Measure: Number; unit: Participants
Arm/Group | Placebo (CP) | Ustekinumab 45 mg (CP)
Number analyzed (Participants) | 162 | 160
Participants | 18 | 132
Statistical Analysis 1: Comparison: Placebo (CP) vs Ustekinumab 45 mg (CP); Null Hypothesis: No difference between ustekinumab 45 mg and placebo for the primary endpoint at a significance level of 0.05. Power calculations were based on two sample size assumptions: 220 (1:1 ratio) and 320 participants (1:1 ratio). Simulation studies evaluated the power to detect a treatment difference between ustekinumab 45 mg group and placebo using a CMH test stratified by baseline weight [<=65 kg vs > 65 kg). The power was >99% for both sample size assumptions; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — The study was designed to maintain a Type I error of 0.05 or less for the primary analysis; Stratified by baseline weight [≤ 65kg vs > 65 kg)]

2. Secondary Outcome: The Number of Patients With a Physician's Global Assessment (PGA) Score of Cleared (0) or Minimal (1) at Week 12
Time Frame: Week 12
Population: All participants were included and analyzed according to their randomized treatment group.
Measure: Number; unit: Participants
Arm/Group | Placebo (CP) | Ustekinumab 45 mg (CP)
Number analyzed (Participants) | 162 | 160
Participants | 24 | 126
Statistical Analysis 1: Comparison: Placebo (CP) vs Ustekinumab 45 mg (CP); Null Hypothesis: No difference between ustekinumab 45 mg and placebo at a significance level of 0.05; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — No multiplicity adjustment was made and nominal p-value was reported; Stratified by baseline weight [≤ 65kg vs > 65 kg)]

3. Secondary Outcome: The Change in Dermatology Life Quality Index (DLQI) From Baseline at Week 12.
Description: Scores could range from 0 to 30. A lower DLQI score represents better quality of life.
Time Frame: Baseline (Week 0) to Week 12
Population: Analysis was based on the subset of participants with evaluable measurements according to their randomized treatment group.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Placebo (CP) | Ustekinumab 45 mg (CP)
Number analyzed (Participants) | 159 | 158
Score | -1.9 (6.63) | -9.3 (7.18)
Statistical Analysis 1: Comparison: Placebo (CP) vs Ustekinumab 45 mg (CP); Null Hypothesis: No difference between ustekinumab 45 mg and placebo at a significance level of 0.05; Test type: Superiority or Other; p < 0.001, ANOVA — No multiplicity adjustment was made and nominal p-value was reported; Analysis of variance on van der Waerden normal scores (Conover, 1980) with treatment and baseline weight (≤ 65kg vs > 65 kg) as factors in the model

ADVERSE EVENTS:
Description: One patient from the 'Placebo (CP)' group was randomized, but never received any treatment. Therefore, he was not included in any safety analysis.
Arm/Group | Placebo (CP) | Ustekinumab 45 mg (CP) | Placebo -> Ustekinumab 45 mg (After CP) | Ustekinumab 45 mg (After CP)
Serious Adverse Events (participants affected / at risk) | 1/161 | 1/160 | 2/158 | 1/159
Other Adverse Events (participants affected / at risk) | 21/161 | 28/160 | 27/158 | 14/159
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (CP) (N=161) | Ustekinumab 45 mg (CP) (N=160) | Placebo -> Ustekinumab 45 mg (After CP) (N=158) | Ustekinumab 45 mg (After CP) (N=159)
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (CP) (N=161) | Ustekinumab 45 mg (CP) (N=160) | Placebo -> Ustekinumab 45 mg (After CP) (N=158) | Ustekinumab 45 mg (After CP) (N=159)
Nasopharyngitis (Infections and infestations) | 13 | 19 | 15 | 7
Upper respiratory tract infection (Infections and infestations) | 8 | 9 | 12 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less